CLINICAL TRIAL: NCT02934295
Title: Study of Rubella Immunity. Response to Vaccination of Subjects With Very Low, Equivocal or Undetectable Titers of Rubella Virus Antibodies
Acronym: ImmRubVac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011/61; 2011-A01445-36 (Other: ANSM)
Record Dates: First submitted 2016-10-13; First posted 2016-10-14 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Pregnancy
Keywords: Rubeola
MeSH Terms: conditions — Measles | interventions — methyl N-acetylsibirosaminide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant women (Experimental)
  Interventions: Biological: Determination of Anti-Rubella Antibody, E1

INTERVENTIONS:
Biological: Determination of Anti-Rubella Antibody, E1

SUMMARY:
The aim of the research is to study humoral and cellular immunity in pregnant women for who the level of rubella virus antibodies is weakly positive, equivocal or negative with the usual laboratory technique.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18
* Rubella serology negative, ambiguous or weakly positive during a first prenatal consultation and for which the second determination of the immunity anti rubella is necessary after 18 weeks of pregnancy
* Accepting the rubella vaccination after the childbirth;
* Accepting a blood test, during a postnatal consultation, 6 in 8 weeks after vaccination, to verify their immunity towards the virus of the rubella.
* Affiliated to a social security scheme
* Having given a written consent

Exclusion Criteria:

* Rubella contracted since the first serology realized during the first prenatal consultation
* Autoimmune pathologies
* Intolerance / allergy known about a previous vaccination whatever it is
* Immunosuppression (HIV, transplants)
* Injection of multivalent immunoglobulins (except anti-D)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Level of Anti-Rubella Antibody, E1 | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Picone, Principal Investigator — Hôpital Foch; Christelle VAULOUP-FELLOUS, MD, Study Chair — Hôpital Brousse
Locations (2):
- France (2):
  - Hôpital Antoine-Béclère, Clamart
  - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No